CLINICAL TRIAL: NCT05736341
Title: Comparison of Remimazolam and Midazolam for Preventing Intraoperative Nausea and Vomiting During Cesarean Section Under Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2022-1528
Record Dates: First submitted 2023-02-01; First posted 2023-02-21 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2023-06

CONDITIONS: Pregnancy; Cesarean Section; Spinal Anesthesia
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam (Experimental): Patient group who receives remimazolam for sedation after delivery
  Interventions: Drug: Remimazolam besylate
- Midazolam (Active Comparator): Patient group who receives midazolam for sedation after delivery
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Remimazolam besylate — After delivery, patients in this group receives 5mg of remimazolam to induce sedation during the remaining procedures of Cesarean section.
  Arms: Remimazolam
Drug: Midazolam — After delivery, patients in this group receives 2mg of midazolam to induce sedation during the remaining procedures of Cesarean section.
  Arms: Midazolam

SUMMARY:
Spinal anesthesia is widely accepted as the anesthetic method of choice for Cesarean section. However, high-level blockage or hypotension induced by this technique may induce intraoperative nausea and vomiting (IONV), which is associated with patient discomfort and protrusion of abdominal viscera which may adversely affect patient safety. To prevent IONV, midazolam is frequently administered after delivery, but risk of hypotension and prolonged sedation due to its active metabolite also increases. On the other hand, remimazolam is known to have relatively shorter half-life and less likely induce hypotension when compared to midazolam, yet its effect on IONV has not been thoroughly evaluated. Hence, this study aimed to compare the effects of remimazolam and midazolam in preventing IONV in patients scheduled for elective Cesarean section.

ELIGIBILITY:
Inclusion Criteria:

Patients (age ≥ 20yrs and ASA Class II or III) who are scheduled for elective Cesarean section

Exclusion Criteria:

Emergency surgery Patients who are diagnosed preeclampsia or eclampsia, BMI ≥ 40kg/m2, IUP < 36 weeks Patients with contraindications to spinal anesthesia Patients who do not want sedation during the procedure

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — As this study evaluates intraoperative nausea and vomiting during Cesarean section, only female participants are eligible to this study.
Enrollment: 80 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2024-01-06 (Actual)

PRIMARY OUTCOMES:
intraoperative nausea and vomiting during sedative period | at 5 minutes after sedative administration
  Incidence of intraoperative nausea, retching, and vomiting will be evaluated 5, 10, 15, 20, 25, 30, and 60 minutes after sedative administration, and at the end of surgery.
intraoperative nausea and vomiting during sedative period | at 10 minutes after sedative administration
  Incidence of intraoperative nausea, retching, and vomiting will be evaluated 5, 10, 15, 20, 25, 30, and 60 minutes after sedative administration, and at the end of surgery.
intraoperative nausea and vomiting during sedative period | at 15 minutes after sedative administration
  Incidence of intraoperative nausea, retching, and vomiting will be evaluated 5, 10, 15, 20, 25, 30, and 60 minutes after sedative administration, and at the end of surgery.
intraoperative nausea and vomiting during sedative period | at 20 minutes after sedative administration
  Incidence of intraoperative nausea, retching, and vomiting will be evaluated 5, 10, 15, 20, 25, 30, and 60 minutes after sedative administration, and at the end of surgery.
intraoperative nausea and vomiting during sedative period | at 25 minutes after sedative administration
  Incidence of intraoperative nausea, retching, and vomiting will be evaluated 5, 10, 15, 20, 25, 30, and 60 minutes after sedative administration, and at the end of surgery.
intraoperative nausea and vomiting during sedative period | at 30 minutes after sedative administration
  Incidence of intraoperative nausea, retching, and vomiting will be evaluated 5, 10, 15, 20, 25, 30, and 60 minutes after sedative administration, and at the end of surgery.
intraoperative nausea and vomiting during sedative period | at 60 minutes after sedative administration
  Incidence of intraoperative nausea, retching, and vomiting will be evaluated 5, 10, 15, 20, 25, 30, and 60 minutes after sedative administration, and at the end of surgery.
intraoperative nausea and vomiting during sedative period | at the end of surgery
  Incidence of intraoperative nausea, retching, and vomiting will be evaluated 5, 10, 15, 20, 25, 30, and 60 minutes after sedative administration, and at the end of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Seung Hyun Kim, Principal Investigator — Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Severance Hospital, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea